CLINICAL TRIAL: NCT02307396
Title: Evaluation of the Necessity of Long-term Pharmacological Treatment With Antipsychotics for the Prevention of Relapse in Long-term Stabilized Schizophrenic Patients: a Randomized, Single-blind, Longitudinal Trial
Brief Title: Evaluation of the Necessity of Long-term Pharmacological Treatment With Antipsychotics in Schizophrenic Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1723/1-1; 2013-000338-37 (EudraCT Number); DO 1723/1-1 (Other Grant/Funding Number: DFG (Deutsche Forschungs Gesellschaft)); DRKS00006878 (Other: Deutsches Register Klinischer Studien)
Record Dates: First submitted 2014-11-24; First posted 2014-12-04 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Schizophrenia; Schizophrenia and Disorders With Psychotic Features; Schizoaffective Disorders
MeSH Terms: conditions — Schizophrenia; Schizophrenia Spectrum and Other Psychotic Disorders; Psychotic Disorders | interventions — Olanzapine; Amisulpride; Risperidone; Haloperidol; Quetiapine Fumarate; Perphenazine; Sulpiride; bromperidol; Clopenthixol; Thioridazine; Paliperidone Palmitate; ziprasidone; Benperidol; Fluspirilene; Pimozide; Perazine; Fluphenazine; sertindole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Intervention group: guided discontinuation or dose-reduction of the current antipsychotic medication. The antipsychotic drug used before study start will be discontinued gradually under medical surveillance. The process of discontinuation depends on the physicians judgement und should be guided be the participants needs and clinical status. This approach was already used before in another study ("gradual discontinuation", Wunderink et al., 2007). We assume that the dose can be reduced by approximately 1/6 of the starting dose every two weeks. If long acting antipsychotics are applied, there is no need for a gradual discontinuation due to their long half life.
  Interventions: Drug: Olanzapine; Drug: Amisulpride; Drug: Risperidone; Drug: Haloperidol; Drug: Quetiapine; Drug: Perphenazine; Drug: Sulpiride; Drug: bromperidol; Drug: Zuclopenthixol; Drug: Thioridazine; Drug: Paliperidone; Drug: Ziprasidone; Drug: Benperidol; Drug: Fluspirilene; Drug: Pimozide; Drug: Perazine; Drug: Fluphenazine; Drug: Flupentixole; Drug: Sertindole
- Control (Active Comparator): The participants receive the same antipsychotic drugs, they have received before the start of the study, without changing the dose or the application form. Study medication is, with exception of Clozapin, every oral or depot neuroleptic drug approved for the treatment of schizophrenia in Germany.
  Interventions: Drug: Olanzapine; Drug: Amisulpride; Drug: Risperidone; Drug: Haloperidol; Drug: Quetiapine; Drug: Perphenazine; Drug: Sulpiride; Drug: bromperidol; Drug: Zuclopenthixol; Drug: Thioridazine; Drug: Paliperidone; Drug: Ziprasidone; Drug: Benperidol; Drug: Fluspirilene; Drug: Pimozide; Drug: Perazine; Drug: Fluphenazine; Drug: Flupentixole; Drug: Sertindole

INTERVENTIONS:
Drug: Olanzapine
Drug: Amisulpride
Drug: Risperidone
Drug: Haloperidol
Drug: Quetiapine
Drug: Perphenazine
Drug: Sulpiride
Drug: bromperidol
Drug: Zuclopenthixol
Drug: Thioridazine
Drug: Paliperidone
Drug: Ziprasidone
Drug: Benperidol
Drug: Fluspirilene
Drug: Pimozide
Drug: Perazine
Drug: Fluphenazine
Drug: Flupentixole
Drug: Sertindole

SUMMARY:
The main objective of the trial is to evaluate, how long an antipsychotic relapse-prevention should be continued and to which time a patient with schizophrenia is protected enough, so that a withdrawal or reduction of the medication seems appropriate. Relapse is defined as primary outcome.

DETAILED DESCRIPTION:
The main objective of the trial is to evaluate for the first time, how long an antipsychotic relapse-prevention should be continued and to which time a patient is protected enough, so that a guided withdrawal or reduction of the medication seems appropriate. Relapse is defined as primary outcome. We include patients with schizophrenia or schizoaffective disorder in remission for at least 3 years under a stable antipsychotic medication.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia or schizoaffective disorder
* The participants have to be in remission for at least 3 years (i.e. no psychiatric hospitalisation) under a stable antipsychotic medication. Remission will be measured using the remission criteria by Andreasen et al. (2005) Score ≤3 for the items concerning psychosis of the "Positive and Negative Syndrom Scale" (PANSS; Kay et al., 1987): "Delusions" (P1), "Conceptual disorganisation" (P2), "Halluzinations" (P3), "Mannerisms and posturing" (G5) and "Unusual thought content" (G9) and a score ≤3 on the "Clinical Global Impression Severity Scale" (CGI-S; Guy, 1976)
* Able to give informed consent

Exclusion Criteria:

* Actively suicidal
* Serious medical illnesses
* Known non-complience concerning the medication
* Medication with clozapin
* Medication with antidepressants and mood stabilisors that were initiated during the last 6 weeks before study enrollment
* Patients with substance dependence other than nicotine or caffeine within 6 months prior to baseline
* Unability to give informed consent
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

PRIMARY OUTCOMES:
Relapse | Every 2 weeks up to 26 weeks
  The criterion is measured at every visit (every two weeks) two weeks with two criteria, both have to be fullfilled:
  1. Score ≥4 (moderate) for at least two of the following PANSS-items :
     "Delusions" (P1), "Conceptual disorganisation" (P2), "Halluzinations" (P3), "Mannerisms and posturing" (G5) and "Unusual thought content" (G9) (PANSS; Kay et al., 1987)
  2. Score ≥4 on the "Clinical Global Impression Severity Scale" (CGI-S; Guy, 1976b)

SECONDARY OUTCOMES:
Psychiatric rehospitalisation | Every 2 weeks up to 26 weeks
Totalscore of Positive and Negative Syndrome Scale (PANSS) | Baseline, then every 4 weeks up to 26 weeks
  PANSS-Scale
Occurence of specific adverse effects (open interview) | Baseline,then every 4 weeks up to 26 weeks
Clinical Global Impression - Severity Scale (CGI-S) | Baseline, then every 4 weeks up to 26 weeks
  CGI-I Scale
"Quality of life" measured by the questionnaire "Subjective well-being under neuroleptics scale" (SW-N) | Baseline, and after 12 and 26 weeks
  SW-N-Scale
Status of occupation | Baseline, and after 12 and 26 weeks
Personal and Social Performance (Personal and Social Performance Scale [PSP]) | Baseline, and after 12 and 26 weeks
  PSP-Scale
Adherence/Attitude of patients towards medication (Medication Adherence Rating Scale [MARS]) | Baseline, and after 12 and 26 weeks
  MARS-Scale
Drop-outs total and due to specific reasons | Every 2 weeks up to 26 weeks
Movement disorders (Abnormal Involuntary Movement Scale [AIMS]) | Baseline, and after 12 and 26 weeks
  AIMS-Scale
Weight change | Baseline, and after 12 and 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Leucht, Professor, Principal Investigator — Klinikum rechts der Isar; Markus Dold, MD, Principal Investigator — Klinikum rechts der Isar
Locations (1):
- Psychiatrische Klinik und Poliklinik fuer Psychiatrie und Psychotherapie der Technischen Universitaet Muenchen am Klinikum rechts der Isar, Munich, Bavaria, Germany